CLINICAL TRIAL: NCT03072836
Title: Study of Gut Microbiota in Crohn's Disease Patients Suffering From Spondylarthritis
Acronym: FLORACROHN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pr Laurent PEYRIN BIROULET, Professor, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2016-A01720-51
Record Dates: First submitted 2017-03-02; First posted 2017-03-07 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Crohn Disease; Spondyloarthritis
MeSH Terms: conditions — Crohn Disease; Spondylarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CD alone (Experimental)
  Interventions: Other: analysing microbiota
- SPA alone (Experimental)
  Interventions: Other: analysing microbiota
- CD + SPA (Experimental)
  Interventions: Other: analysing microbiota

INTERVENTIONS:
Other: analysing microbiota — 16SRNA gene sequencing of feces

SUMMARY:
The FLORACROHN project aims to compare gut microbiota of patients suffering from Crohn's disease (CD) associated or not to spondylarthritis (SpA).

3 groups of patients will be analyzed: patients suffering from CD alone, patients suffering from SpA alone, patients suffering from CD and SpA.

Fecal microbiota will be determined by 16SRNA gene sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Crohn's disease and axial spondyloarthritis according to the criteria below.

  * Patients with Crohn's disease (CT patients) diagnosed according to clinical, biological, radiological, endoscopic and / or histological criteria for 3 months. With diagnosis of spondyloarthritis exclusion on modified ASAS and / or New York criteria.
  * Patients with axial spondyloarthritis (SpA patients) diagnosed according to the modified ASAS and / or New York criteria with exclusion diagnosis of Crohn's disease.
* Patient with the capacity to give free and informed consent.

Exclusion Criteria:

Antecedent of colonic resection

* Antibiotic or colonic colonoscopy preparation in the 8 weeks prior to stool collection (against temporary indication = collection possible before colic preparation or on the first saddle after the start of the colic preparation).
* Ostomy at time of collection
* BMI> 30
* extreme diet
* unbalanced diabetes
* Patient under guardianship, under curatorship or under safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2017-03-06 (Actual); Primary Completion 2020-05-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Microbiota analysis | 6 months after last patient inclusion
  16SRNA gene sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No